CLINICAL TRIAL: NCT07099651
Title: Ataxies SpinoCérébelleuses Autosomiques Dominantes et Cognition Sociale - Etude SoCoSca
Brief Title: Autosomal Dominant Spinocerebellar Ataxias and Social Cognition
Acronym: SoCoSca
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 49RC23-0390; ID-RCB 2025-A01253-46 (Other: ANSM)
Record Dates: First submitted 2025-07-17; First posted 2025-08-01 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Autosomal Dominant Spinocerebellar Ataxia (SCA1, 2,3,6,7,27B)
MeSH Terms: conditions — Spinocerebellar Ataxias

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- patients autosomal dominant spinocerebellar ataxia (Active Comparator)
  Interventions: Other: tests
- healthy patients (Active Comparator)
  Interventions: Other: tests

INTERVENTIONS:
Other: tests — neuropsychological tests + Neuroimaging

SUMMARY:
Spinocerebellar ataxias are a group of rare neurodegenerative diseases, clinically and genetically highly heterogeneous, with an estimated mean prevalence of 2.7 per 100,000 population. The term "spinocerebellar ataxia" or "SCA" is often used for ataxias of genetic origin of autosomal dominant transmission, which are the subject of this study. Recent studies of social cognition in patients with genetic cerebellar pathologies, and autosomal dominant spinocerebellar ataxia in particular, are still few and far between (around 15 studies), and seem to highlight impairment of basic emotion recognition and theory of mind skills. That said, data have very often been collected on very small samples of patients (sometimes in case study format). They also remain contradictory, including in the examination of the cerebellar anatomoclinical correlates of the deficits. Thus, the question arises as to whether patients with spinocerebellar ataxia also show impairments in emotion recognition and cognitive and affective theory of mind in more ecologically valid dynamic and interactive assessment situations.

ELIGIBILITY:
Inclusion Criteria:

For all participants:

* Men or women aged 18 and over
* At least 7 years' schooling (CEP level)
* Ability to read, write and speak French
* Signed informed consent to participate in the study

For patients :

- With molecularly confirmed autosomal dominant spinocerebellar ataxia (SCA1, 2, 3, 6, 7, 27B)

For controls:

- With no neurological pathology (questioning and neurological examination)

Exclusion Criteria:

For patients and controls:

* Simultaneous participation in another protocol that may interfere with the measurement of the criteria of interest
* Physical or cultural factors likely to interfere with test performance
* History likely to interfere with cognition (stroke, cranioencephalic trauma, other neurodegenerative disease, epilepsy, learning disability, alcohol dependence syndrome, psychiatric disorders...)
* Persons with contraindications to MRI scans
* Pregnant, nursing or parturient women
* Persons deprived of their liberty by judicial or administrative decision
* Persons under compulsory psychiatric care
* Persons subject to a legal protection measure
* Persons unable to express their consent
* Persons not affiliated to or not benefiting from a social security scheme (beneficiary or beneficiary entitled)

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2025-12-09 (Actual); Primary Completion 2028-11-01 (Estimated); Study Completion 2029-01-01 (Estimated)

PRIMARY OUTCOMES:
to assess the social cognition with the Facial Emotion Recognition Test from classical approach | Baseline
  Facial Emotion Recognition Test evaluates the ability to recognize 6 fundamental and universal emotions: happiness, anger, sadness, fear, disgust and contempt. Each emotion is expressed by a different face at 9 levels of expressive intensity, ranging from 20% to 100%
to assess the social cognition with the Faux Pas Test from classical approach | Baseline
  Faux Pas Test: in its shortened 10-story version, it assesses the ability to recognize social awkwardness (or faux-pas). Fictitious stories are presented to the person, in paper format: 5 stories contain faux-pas and 5 others do not. The person can reread them as many times as necessary, and must detect whether "someone said something they shouldn't have, or something awkward". If this is the case, she is asked 5 additional questions to assess her understanding of the clumsiness. Each story is followed by 2 comprehension questions, to rule out a comprehension problem. This task takes 20 minutes to administer. The test produces different scores: the higher the score, the better the performance.
to assess the social cognition with the Reading the Mind in the Eyes test from classical approach | Baseline
  Reading the Mind in the Eyes test: Thirty-six photographs of gazes (male and female) are presented to the participant, who is asked to select from 4 expression proposals the one that seems most appropriate to the subject's affective mental state (what he or she may be feeling). A lexicon that can be consulted at will is provided to the subject to compensate for any uncertainties concerning the proposed items. The maximum score is 36 (1 point per correctly chosen item). The test takes 15 to 20 minutes to complete.
to assess the social cognition with the sequencing test from classical approach | Baseline
  sequencing test: sequential arrangement of 12 scenarios, all consisting of 4 images in the format of short comic strips. They represent mechanical (non-social) events and social scripts including true (4 scenarios) and false beliefs (4 scenarios). Subjects are asked to put each image sequence, presented in random order, back into chronological order. There are 4 non-social scenarios, 4 true-belief scenarios and 4 false-belief scenarios for a 12-point score. The test begins with 2 practice trials. The test lasts 20 minutes.
to assess the social cognition with the French Emotion Evaluation Test from ecological approach | Baseline
  French Emotion Evaluation Test: audiovisual, ecological and valid emotion recognition test. It tests subjects' ability to recognize basic emotions expressed by other people. It comprises 35 short video sequences (15 to 30 seconds) plus an example item. In each of these sequences, actors interpret everyday situations associated with one of the 6 basic emotions: joy, sadness, anger, surprise, disgust and fear. The test produces a total response score of between 0 and 35.
to assess the social cognition with the Movie for the Assessment of Social Cognition Test from ecological approach | Baseline
  evaluates theory of mind in dynamic modality. It was adapted and validated in French (MASC-VF) as part of a partnership between Patricia Garel's team (Hopital Universitaire de Sainte-Justine, Montreal, Quebec) and Isabelle Amado's team (Centre Hospitalier Sainte-Anne, Service Hospitalo-Universitaire, Paris, France). This test assesses both the affective and cognitive sides of theory of mind, and also includes six control questions to rule out a comprehension problem. The test takes around 40 minutes to administer. The test will assess the cognitive and affective theory-of-mind abilities of ALS patients in comparison with those of matched control subjects. The MASC calculates 5 scores: 1 comprehension score, 1 correct response score ranging from 0 to 45 points and 3 error scores (wrong answers are divided into 3 categories: under-interpretation error, over-interpretation error and no interpretation). The higher the score of correct answers, the better the performance.
to assess the social cognition with the social problem-solving test from interactionist approach | Baseline
  This test has been developped at Angers . A total of 10 stories involving social problems will be proposed. For 5 of them, the participant will have to produce verbal solutions, and for the other 5, act them out in a social role-playing situation, with a partner. The test lasts 40 minutes.

SECONDARY OUTCOMES:
Search for and describe any deficits in social cognition by identifying pathological treshold with Facial Emotion Recognition Test | Baseline
  this test evaluates the ability to recognize 6 fundamental and universal emotions: happiness, anger, sadness, fear, disgust and contempt. Each emotion is expressed by a different face at 9 levels of expressive intensity, ranging from 20% to 100%.
Research and describe any deficits in social cognition by identifying pathological treshold with false step test | Baseline
  it assesses the ability to recognize social awkwardness (or faux-pas). Fictitious stories are presented to the person, in paper format: 5 stories contain faux-pas and 5 others do not. The person can reread them as many times as necessary, and must detect whether "someone said something they shouldn't have, or something awkward". If this is the case, she is asked 5 additional questions to assess her understanding of the clumsiness. Each story is followed by 2 comprehension questions, to rule out a comprehension problem. This task takes 20 minutes to administer. The test yields different scores: the higher the scores, the better the performance.
Research and describe any deficits in social cognition by identifying pathological treshold with Reading the Mind in the Eyes test | Baseline
  Thirty-six photographs of gazes (male and female) are presented to the participant, who is asked to select from 4 expression proposals the one that seems most appropriate to the subject's affective mental state (what he or she may be feeling). A lexicon, which can be consulted at will, is provided to the subject, to compensate for any uncertainties concerning the proposed items. The maximum score is 36 (1 point per correctly chosen item). The test takes 15 to 20 minutes to complete.
Search for and describe any deficits in social cognition by identifying pathological treshold with sequencing test | Baseline
  Subjects must put each image sequence, presented in random order, back into chronological order. There are 4 non-social scenarios, 4 true-belief scenarios and 4 false-belief scenarios for a 12-point score. The test begins with 2 practice trials. The test lasts 20 minutes.
Research and describe any deficits in social cognition by identifying pathological treshold with French Emotion Evaluation Test | Baseline
  This is an audiovisual, ecological and valid emotion recognition test. It tests subjects' ability to recognize basic emotions expressed by other people. It comprises 35 short video sequences (15 to 30 seconds) plus an example item. In each of these sequences, actors interpret everyday situations associated with one of the 6 basic emotions: joy, sadness, anger, surprise, disgust and fear. This task takes 20 minutes to administer. The test yields a total response score of between 0 and 35.
Research and describe any deficits in social cognition by identifying pathological treshold with Movie for the Assessment of Social Cognition | Baseline
  subject watches a 25-minute video featuring four young people meeting on a Saturday night. The video is broken down into 46 scenes. It is interrupted 45 times. Each time, a question is asked about mental states (what does a character feel/think, or what is their intention?). The person being evaluated is then given a choice of four responses, to be situated on a gradient ranging from a literal response (no theory of mind) to an over-interpretive response (too much theory of mind), via a response involving too little theory of mind to the correct response. The MASC calculates 5 scores: 1 comprehension score, 1 correct answers score ranging from 0 to 45 points and 3 error scores (wrong answers are divided into 3 categories: under-interpretation error, over-interpretation error and no interpretation). The higher the score of correct answers, the better the performance.
Research and describe any deficits in social cognition by identifying pathological treshold with social problem-solving test | Baseline
  the participant must describe an interpersonal social problem, find a solution to this problem and/or implement this solution in a simulation with another person (cognitive TDE). This task also includes questions about feelings/emotions in these problem situations, thus assessing the affective component of TDE. A total of 10 stories involving social problems will be proposed. For 5 of them, the participant will have to produce verbal solutions, and for the other 5, act them out in a social role-playing situation, with a partner. The test lasts 40 minutes.
Research and describe any deficits in social cognition by identifying pathological treshold with brain neuroimaging | 3 months
  magnetic resonance imaging
Study correlations between social cognition efficiency and - Global cognitive functioning assessed by the CCAS-S scale | Baseline
  This is a 10-subscale screening measure assessing attention and concentration, executive functioning, memory, language, visuospatial functioning, abstract thinking and major neuropsychiatric features. Each subscale is associated with a raw score and a pass/fail evaluation. The total raw score is a maximum of 120, and the total number of "failed" items is a maximum of 10. The test takes 15 to 20 minutes to complete.
Study correlations between social cognition efficiency and Sociobehavioral and emotional abilities assessed by the Neuropsychiatric Inventory Questionnaire | Baseline
  It assesses 12 different types of behavior (delusions, hallucinations, agitation, depression, anxiety, euphoria, apathy, disinhibition, irritability, aberrant motor behaviors, sleep disorders, appetite disorders). It is based on the responses of an informed caregiver, preferably living with the patient. The severity and frequency of behavioral problems, and their impact on the caregiver, are listed. It can also be completed directly with the patient. Patients are asked to fill in the questionnaire (self- and hetero-assessment), together with their relative if applicable. The questionnaire takes 10 to 15 minutes to complete.
Study correlations between social cognition efficiency and Sociobehavioral and Sociobehavioral and emotional abilities assessed by the Frontal System Behaviour Scale | Baseline
  Items are scored on a 5-point scale: 1 (almost never), 2 (rarely), 3 (sometimes), 4 (often), 5 (almost always). Four scores are obtained: Total, Apathy, Disinhibition and Executive. Scores above T = 65 are considered clinically significant. The test lasts 10 minutes.
Study correlations between social cognition efficiency and Sociobehavioral and Sociobehavioral by Hospital Anxiety and Depression scale | Baseline
  The test takes 10 minutes to complete. It comprises 14 items, rated from 0 to 3. Seven questions relate to anxiety and 7 to depression, giving 2 scores:
  * An anxiety score between 0 and 21. The higher the score, the greater the presence of the disorder.
  * A depression score between 0 and 21. The higher the score, the more the disorder is present.
Study correlations between social cognition efficiency and Sociobehavioral and Sociobehavioral by Ambiguous Intentions Hostility Questionnaire-Short | Baseline
  It assesses the spontaneous attribution of intentions (particularly hostile intentions), the emotion felt and the behavioural response to ambiguous social situations.
  Participants are asked to read each situation and imagine themselves in it. They are then asked to answer several questions to measure three scores: [1] a hostility bias, reflecting the degree of hostility they attribute to the other person's actions towards themselves; [2] a responsibility attribution score, which is the average of three evaluations on Likert scales : an intentionality score (whether the person acted intentionally); an anger score (how angry they would feel) and a blame score (how much they would blame the other person); [3] an aggression bias corresponding to the level of aggression in their response. The questionnaire lasts 20 minutes.
Study correlations between social cognition efficiency and Sociobehavioral and Sociobehavioral by Social Cognitive Impairment Rating Scale | Baseline
  This enables 5 scores to be calculated: a total score out of 48 points and 4 sub-scores out of 12 points corresponding to each area. The questionnaire takes 20 minutes to complete. Patients and their relatives, if applicable, are asked to complete the questionnaire (self- and hetero-assessment).
Study correlations between social cognition efficiency and Sociobehavioral and Sociobehavioral by Bermond-Vorst Alexithymia Questionnaire | Baseline
  This is a self-questionnaire (5-point Likert scale) that measures 5 dimensions: (1) difficulty identifying emotional states The total score is between 20 and 100. The questionnaire takes 5 to 10 minutes to complete.
Study correlations between social cognition efficiency and Sociobehavioral and Sociobehavioral by scale of levels of emotional awareness | Baseline
  It assesses the degree of emotional awareness in relation to oneself and others. The PECS-B version includes 20 stories and assesses the participant's ability to describe their own emotions and those of others in each story. The score is between 0 and 100. The questionnaire takes 10 to 20 minutes to complete.
Study correlations between social cognition efficiency and imaging data | 3 months
  magnetic resonance imaging: imaging analysis (structure, functions, connectivities)
Study correlations between social cognition efficiency and duration of disease progression | Baseline
  duration in months of disease progression
Study correlations between social cognition efficiency and ataxia severity by the Scale for the Assessment and Rating of Ataxia | Baseline
  This is a quick and easy-to-use 40-point scale with 8 items assessing walking, posture, sitting position, articulation, finger pursuit, finger/nose test, rapid alternating movements and movement of the heel on the contralateral tibia. The higher the score, the greater the severity of the ataxia. The SARA is a scale initially validated for vascular spinocerebellar ataxia, and lasts around 15 minutes.
Study the correlations between the efficiency of social cognition and the severity of ataxia as assessed by the International Co-operative Ataxia Rating Scale. | Baseline
  This 100-point scale provides a semi-quantitative, compartmentalised assessment of the various symptoms observed in cerebellar syndrome. It comprises 19 items grouped into four subgroups, which allow different functions to be studied, such as posture and disturbances during walking, kinetic functions, speech disorders and oculomotor disorders. The score takes around 30 minutes to complete.
Study the correlations between the efficiency of social cognition and the severity of ataxia as assessed by neurofilament dosage. | Baseline
  recovery of neurofilament assay data
To study the correlations between the efficiency of social cognition and the global motor skills of the upper limb using the Box and Block test (assessing the gross dexterity of the upper limb tested). | Baseline
  This quick and easy test assesses the overall dexterity of the upper limbs. The subject will be seated, with the equipment placed on a height-adjustable shelf. The score expresses the number of cubes that the subject has transported, with one hand only, from one compartment of the box to another in 1 minute. The results are expressed as the number of cubes transported in one minute. The greater the number of cubes transported, the better the overall dexterity of the upper limb tested. The subject is free to choose which hand is used first. This choice will be noted.
To study the correlations between the efficiency of social cognition and the fine motor skills by the Nine Hole Peg Test | Baseline
  The subject must place 9 pegs in the holes provided. The time taken to put the pegs in and then remove them will be measured. This test is timed. The examiner will explain the task and give a demonstration. The final score in seconds for this test will be used to determine which hand is the most skilful for the fine motor tasks. This assessment will also be carried out on controls. This assessment, carried out routinely for patients followed in Angers, lasts less than 5 minutes.
Study the supposed differences between SCA subtypes, by comparing pure cerebellar forms with cerebro-cerebellar forms and by comparing the different genetic subtypes with each other, using Facial Emotion Recognition Test | Baseline
  assesses the ability to recognise 6 fundamental and universal emotions: happiness, anger, sadness, fear, disgust and contempt. Each emotion is expressed by a different face in 9 levels of expressive intensity ranging from 20 to 100%.
Study the supposed differences between SCA subtypes, by comparing pure cerebellar forms with cerebro-cerebellar forms and by comparing the different genetic subtypes with each other, using False Step Test | Baseline
  .This task takes 20 minutes to administer. The test produces different scores: the higher the scores, the better the performance.
  * Stories containing a misstep :
  * Correct detections: /5 (number of stories containing a misstep for which the subject answered 'yes' to question 1)
  * Total misstep score: /30 (correct detection score above + the sum of the correct answers obtained to questions 2 to 6)
  * Score for the cognitive theory of mind question (Question 5): /5
  * Score for the affective theory of mind question (Question 6): /5
  * Comprehension: /10 (sum of correct answers to questions 7 and 8)
  * Stories containing no errors
  * Correct rejections: /4 (number of stories without errors for which the subject answered 'no' to question 1)
  * Comprehension: /8 (sum of correct answers to questions 7 and 8)
Study the supposed differences between SCA subtypes, by comparing pure cerebellar forms with cerebro-cerebellar forms and by comparing the different genetic subtypes with each other, using Reading the Mind in the Eyes test | Baseline
  Thirty-six photographs of gazes (male and female) are presented to the participant, who is asked to select from 4 suggested expressions the one that seems most appropriate to the subject's affective mental state (what he or she may be feeling). A lexicon that can be consulted at leisure is provided to the subject to compensate for any uncertainties concerning the proposed items. The maximum score is 36 (1 point per correctly chosen item). The test takes 15 to 20 minutes.
Study the supposed differences between SCA subtypes, by comparing pure cerebellar forms with cerebro-cerebellar forms and by comparing the different genetic subtypes with each other, using Sequencing test | Baseline
  Subjects have to put each image sequence, presented in random order, back into chronological order. There are 4 non-social scenarios, 4 true belief scenarios and 4 false belief scenarios for a score out of 12 points. The test begins with 2 practice trials. The test lasts 20 minutes.
Study the supposed differences between SCA subtypes, by comparing pure cerebellar forms with cerebro-cerebellar forms and by comparing the different genetic subtypes with each other, using French Emotion Evaluation Test | Baseline
  After viewing each scene, the test subject chooses the emotion perceived from a list provided, which includes the 6 basic emotions and the 'neutral emotion'. The possible answers are presented in a random order, which changes with each scene. There are 5 response cards. The task takes 20 minutes to administer. The test produces a total response score of between 0 and 35, as well as different sub-scores (correct responses per emotion, correct responses for positive emotions and correct responses for negative emotions). A score on the recognition of the gender of the person photographed is collected to ensure that there is no perceptual disorder. The higher the score, the better the performance.
Study the supposed differences between SCA subtypes, by comparing pure cerebellar forms with cerebro-cerebellar forms and by comparing the different genetic subtypes with each other, using Movie for the Assessment of Social Cognition | Baseline
  The viewer watches a 25-minute video of four young people getting together on a Saturday night. The video is broken down into 46 scenes. It is interrupted 45 times. Each time a question is asked about mental states (what is the character feeling/thinking or what is their intention?). The person being assessed is then given a choice of four responses to be placed on a gradient ranging from a literal response (no theory of mind) to an over-interpretive response (too much theory of mind), via a response that does not involve enough theory of mind and the correct response.
  It calculates 5 scores: 1 comprehension score, 1 correct response score of between 0 and 45 points and 3 error scores (incorrect responses are divided into 3 categories: under-interpretation error, over-interpretation error and no interpretation). The higher the score of correct answers, the better the performance.
Study the supposed differences between SCA subtypes, by comparing pure cerebellar forms with cerebro-cerebellar forms and by comparing the different genetic subtypes with each other, using social problem-solving test | Baseline
  A total of 10 stories about social problems will be proposed. For 5 of them, the participant will have to produce verbal solutions and for the other 5, act them out in a social interaction situation with a partner. The test lasts 40 minutes.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Angers, Angers, France

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared upon reasonable request. Only de-identified data will be shared. Any data collected during the study may be shared. The protocol will be shared initially. Other documents may be shared at a later date upon request (e.g., the CRF to allow a collaborator to select the data they wish to access). The recipients of the data will be researchers. The data will be available for any purpose deemed relevant by the study investigator, based on a protocol provided by the requester, after verification of the obtaining of regulatory approvals, including the favorable opinion of an ethics committee.
Supporting Information: Study Protocol
Time Frame: The data will be shared after signing a negotiated data transfer agreement ( data access agreement), for the duration specified in the agreement.
Access Criteria: The data will be made available via secure transfer (sharing platform approved by the university hospital: BlueFiles or Oodrive).